CLINICAL TRIAL: NCT06052228
Title: Cultural Adaptation and Turkish Version of the Worry About Pain Questionnaire in Individuals With Musculoskeletal Pain: Reliability and Validity Study
Brief Title: Turkish Version of the Worry About Pain Questionnaire
Status: Completed | Type: Observational
Sponsor: Istinye University (Other)
Responsible Party: Principal Investigator, Kubra Koce, Lecturer, Istinye University
Other Study IDs: 21-39
Record Dates: First submitted 2023-09-18; First posted 2023-09-25 (Actual); Last update posted 2024-02-21 (Actual); Status verified 2024-02

CONDITIONS: Pain, Chronic; Musculoskeletal Pain
MeSH Terms: conditions — Chronic Pain; Musculoskeletal Pain

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Assessment Group: Evaluation forms will be applied to the participant who meets the inclusion criteria by face-to-face interview method. The sociodemographic information of the participants and the time taken to answer the questions in the questionnaires will vary according to each participants but will take approximately 45 minutes. The second interview will be conducted with the patients for test-retest application at 1-week intervals.
  Interventions: Other: Assessment Group

INTERVENTIONS:
Other: Assessment Group — Evaluation forms will be applied to the participant who meets the inclusion criteria by face-to-face interview method. The sociodemographic information of the participants and the time taken to answer the questions in the questionnaires will vary according to each participants but will take approximately 45 minutes. The second interview will be conducted with the patients for test-retest application at 1-week intervals.

SUMMARY:
Pain is one of the main complaints that causes people to apply to health institutions. Pain is seen as a passive warning signal of an underlying disease process; When it becomes chronic, it is considered a disease on its own. Pain that persists longer than the expected recovery time is defined as chronic pain.

Pain is associated with a number of psychological, physical, and social factors. Clinical observations report that various psychological problems, especially anxiety, and depression, accompany chronic pain, and the long-term persistence of pain significantly impacts a patient's quality of life. Chronic musculoskeletal pain causes fatigue, sleep disruption, and activity and participation restrictions. Therefore, evaluation of pain originating from the musculoskeletal system and factors that cause and increase pain need to be addressed from a biopsychosocial perspective. Chronic pain is an ideal environment for anxiety to develop. If the person's chronic pain cannot be resolved, anxiety increases and the anxiety becomes excessive, the person may lose the ability to distinguish what is dangerous from what is not, as he cannot evaluate pain-related cues properly. Anxiety and depression scales are often used to assess the long-term psychosocial consequences of chronic musculoskeletal pain. However, these scales are inadequate to explain the relationship between pain and anxiety. The Worry About Pain Questionnaire is a self-report scale of 15 items specifically developed to assess pain-related pressure.

To our knowledge, there is no standard, valid, and reliable Turkish questionnaire in the literature that evaluates the pain-related concerns of individuals with musculoskeletal pain and takes into account the cultural differences of Turkish patients. For this reason, our study aims to translate and culturally adapt the Worry About Pain Questionnaire into Turkish in individuals with chronic musculoskeletal pain and to examine the psychometric properties of the Turkish Worry About Pain Questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* Being able to read and write in Turkish
* Not having any cognitive impairment
* Having chronic musculoskeletal pain
* Being over 18 years of age
* Being willing and volunteer to work

Exclusion Criteria:

* Having a complaint of pain in the musculoskeletal system due to cancer, fracture or surgery within the last 6 months.
* Having severe cognitive impairment
* Having a systemic disease such as rheumatoid arthritis, diabetes mellitus
* Having any neuromuscular disease (such as MS, myopathy)

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Individuals with Musculoskeletal Pain
Sampling Method: Probability Sample
Enrollment: 85 (Actual)
Dates: Start 2023-11-20 (Actual); Primary Completion 2024-02-01 (Actual); Study Completion 2024-02-20 (Actual)

PRIMARY OUTCOMES:
The Worry About Pain Questionnaire | 4 weeks
  The Worry About Pain Questionnaire will be used to evaluate participants' pain-related anxiety levels. Worry About Pain Questionnaire is a Likert-type survey consisting of a total of 15 items. Each question in the survey is scored from 0 (never) to 10 (always). Questions 1, 2, 4, 5, 6, 7, 8, 10, 11, 12 assess the impact of worrying about pain. Questions 3, 9, 13, 14, 15 assess concern about the ability to manage pain.
Fear of Pain Scale III | 4 weeks
  Fear of Pain Scale III, which is used to evaluate the participants' fear of pain, consists of a total of 30 items. A Turkish validity and reliability study was conducted by Ünver et al. in 2018.
Short Form McGill Pain Scale | 4 weeks
  The McGill Pain Scale Short Form combines the features of the standard McGill Pain Questionnaire and is used to evaluate pain caused by chronic cancer pain, chronic back pain, fibromyalgia syndrome, osteoarthritis pain, neuropathic pain, mastalgia and rheumatoid arthritis. Turkish validity and reliability study was conducted by Yakut et al. in 2007.
Pain Pressure Threshold | 4 weeks
  Pressure algometer (dolorimeter) will be used to evaluate sensitivity to pain and determine pressure perception. Pressure algometers have proven useful in assessing fibrositis and hypersensitive points, trigger points, arthritis activation, and visceral pain-pressure sensitivity. For this reason, in our study, the pain pressure threshold will be determined from the trigger points in the upper, middle and lower fibers of the trapezius muscle.

SECONDARY OUTCOMES:
Beck Depression Inventory, | 4 weeks
  Beck Depression Inventory, which is among the most used scales to measure depression all over the world, consists of a total of 21 questions. Each item receives points between 0-3. 11-17 points indicate mild depression, 18-29 points indicate moderate depression, and 30-63 points indicate severe depression. The scale is one of the most widely used depression scales in clinics in Turkey.
Beck Anxiety Inventory | 4 weeks
  Beck Anxiety Inventory, which is used to evaluate the anxiety symptoms experienced by individuals due to social isolation, consists of 21 items and is scored between 0-3. 0-21 points indicate low anxiety, 22-35 points indicate moderate anxiety, and 36 points and above indicate high anxiety.
Nottingham Health Profile | 4 weeks
  The Nottingham Health Profile was developed in England in 1985 to evaluate the health-related quality of life in individuals and has been translated into many languages. The Nottingham Health Profile is a general quality of life survey that evaluates individuals' health problems and the extent to which the problems affect their daily living activities. In 2000, its Turkish validity and reliability were tested in patients with osteoarthritis by Küçükdeveci et al. Nottingham Health Profile Survey consists of a total of 38 questions and 6 subheadings. Subheadings were classified as energy (3 items), social isolation (5 items), pain (8 items), sleep (5 items), physical activity (8 items) and emotional reactions (9 items). The answers to the questions are defined as Yes/No. Each subheading is scored between 0-100. A high total score indicates poor health status.
Pittsburgh Sleep Quality Index | 4 weeks
  Pittsburgh Sleep Quality Index is a scale that provides information about sleep quality and the type and severity of sleep disturbance in the last month. In this scale, the person's sleep quality; Sleep latency is evaluated by sleep duration, habitual sleep efficiency, sleep disturbance, use of sleeping pills, and daytime dysfunction. The Turkish validity and reliability study of the scale was conducted by Ağargün et al. Each survey question is given a score of 0-3, with higher scores reflecting poor sleep quality. If the total score obtained from the scale is less than 5, it is defined as 'Good sleep quality', and if it is 5 or above, it is defined as 'Bad sleep quality'.
Tampa Kinesiophobia Scale | 4 weeks
  Tampa Kinesiophobia Scale is a 17-question scale developed to measure the fear of movement/re-injury. The scale includes injury/re-injury and fear-avoidance parameters in work-related activities. A Turkish validity and reliability study was conducted by Yılmaz et al. in 2011.

CONTACTS AND LOCATIONS:
Locations (1):
- Istinye University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No